CLINICAL TRIAL: NCT02753413
Title: An Observer-blind Safety and Reactogenicity Study to Assess GlaxoSmithKline (GSK) Biologicals' Investigational Respiratory Syncytial Virus (RSV) Vaccine (GSK3003891A) in Healthy Women
Brief Title: Safety and Reactogenicity Study of GlaxoSmithKline (GSK) Biologicals' Investigational Respiratory Syncytial Virus (RSV) Vaccine (GSK3003891A) in Healthy Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 204813; 2015-005742-58 (EudraCT Number)
Record Dates: First submitted 2016-04-21; First posted 2016-04-27 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Vaccine; Safety; Reactogenicity; Respiratory syncytial virus (RSV)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- RSV group (Experimental): Subjects in this group will receive a single dose of the RSV vaccine.
  Interventions: Biological: RSV vaccine GSK3003891A
- Boostrix group (Active Comparator): Subjects in this group will receive a single dose of Boostrix.
  Interventions: Biological: Boostrix

INTERVENTIONS:
Biological: RSV vaccine GSK3003891A — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm.
  Arms: RSV group
Biological: Boostrix — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm.
  Arms: Boostrix group

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of a single intramuscular dose of GSK Biologicals' investigational RSV vaccine, in healthy, non-pregnant women aged 18 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* Non-pregnant female between, and including, 18 and 45 years of age at the time of vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception during the entire study period.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days prior to study vaccination, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Chronic administration of immunosuppressants or other immune-modifying drugs, as well as administration of long-acting immune-modifying drugs during the period starting 6 months prior to study vaccination, or planned administration during the study period. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before study vaccination or planned administration during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the study vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before or after study vaccination.
* Previous experimental vaccination against RSV.
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of or current auto-immune disease.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality as determined by physical examination and/or Medical History.
* Lymphoproliferative disorder or malignancy within previous 5 years.
* History of hypersensitivity after a previous dose of any tetanus, diphtheria, or pertussis vaccine or to any component of Boostrix.
* History of encephalopathy of unknown aetiology occurring within 7 days following a previous vaccination with pertussis-containing vaccine.
* History of any neurological disorders or seizures.
* History of transient thrombocytopenia or neurological complications following a previous vaccination against diphtheria and/or tetanus.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccines.
* Hypersensitivity to latex.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Current chronic alcohol consumption and/or drug abuse.
* Acute disease and/or fever at the time of enrolment.
* Body mass index (BMI) > 40 kg/m2.
* Pregnant or lactating female.
* Planned move to a location that will prohibit participating in the trial until study end.
* Any other condition that the investigator judges may interfere with study procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-04-01; Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Beran J, Lickliter JD, Schwarz TF, Johnson C, Chu L, Domachowske JB, Van Damme P, Withanage K, Fissette LA, David MP, Maleux K, Schmidt AC, Picciolato M, Dieussaert I. Safety and Immunogenicity of 3 Formulations of an Investigational Respiratory Syncytial Virus Vaccine in Nonpregnant Women: Results From 2 Phase 2 Trials. J Infect Dis. 2018 Apr 23;217(10):1616-1625. doi: 10.1093/infdis/jiy065. PMID 29401325
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 102 subject numbers were screened, but only 100 subjects were randomized and received vaccination.
Groups:
- GSK3003891A Group: Healthy, non-pregnant women, aged 18-45 at the time of vaccination, were administered one dose of the investigational GSK3003891A vaccine, intramuscularly in the deltoid region of the arm, at Day 0
- Boostrix Group: Healthy, non-pregnant women, aged 18-45 at the time of vaccination, were administered one dose of the comparator Boostrix™ vaccine, intramuscularly in the deltoid region of the arm, at Day 0
Period: Overall Study
Arm/Group | GSK3003891A Group | Boostrix Group
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3003891A Group | Boostrix Group | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.80 (5.90) | 25.60 (6.10) | 25.70 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Abnormal Biochemical Laboratory Values.
Description: Among analysed biochemical parameters were alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine [CRE]. Biochemical value ranges assessed were below, within or above, as compared to baseline at Day 0.
Time Frame: At Day 7
Population: The analysis was performed on the Total Vaccinated Cohort (TVC) which included all subjects with study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  ALT, Within-Bellow | 0 | 0
  ALT, Within-Within | 48 | 50
  ALT, Within-Above | 1 | 1
  AST, Within-Below: number analyzed (Participants) | 48 | 51
  AST, Within-Below | 0 | 0
  AST, Within-Within: number analyzed (Participants) | 48 | 51
  AST, Within-Within | 48 | 48
  AST, Within-Above: number analyzed (Participants) | 48 | 51
  AST, Within-Above | 0 | 3
  AST, Above-Below: number analyzed (Participants) | 1 | 0
  AST, Above-Below | 0 | 0
  AST, Above-Within: number analyzed (Participants) | 1 | 0
  AST, Above-Within | 0 | 0
  AST, Above-Above: number analyzed (Participants) | 1 | 0
  AST, Above-Above | 1 | 0
  CRE, Within-Bellow | 0 | 0
  CRE, Within-Within | 49 | 51
  CRE, Within-Above | 0 | 0

2. Primary Outcome: Number of Subjects With Abnormal Biochemical Laboratory Values.
Description: as for outcome 1
Time Frame: At Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  ALT, Within-Bellow | 0 | 0
  ALT, Within-Within | 48 | 51
  ALT, Within-Above | 1 | 0
  AST, Within-Below: number analyzed (Participants) | 48 | 51
  AST, Within-Below | 0 | 0
  AST, Within-Within: number analyzed (Participants) | 48 | 51
  AST, Within-Within | 47 | 51
  AST, Within-Above: number analyzed (Participants) | 48 | 51
  AST, Within-Above | 1 | 0
  AST, Above-Below: number analyzed (Participants) | 1 | 0
  AST, Above-Below | 0 | 0
  AST, Above-Within: number analyzed (Participants) | 1 | 0
  AST, Above-Within | 0 | 0
  AST, Above-Above: number analyzed (Participants) | 1 | 0
  AST, Above-Above | 1 | 0
  CRE, Within-Bellow | 0 | 0
  CRE, Within-Within | 49 | 51
  CRE, Within-Above | 0 | 0

3. Primary Outcome: Number of Subjects With Abnormal Haematological Laboratory Values.
Description: Among analysed haematological parameters were eosinophils [EOS], haemoglobin [Hgb], leukocytes (white blood cells) [WBC], lymphocytes [LYM], neutrophils [NEU] and platelets [PLT]. Haematological value ranges assessed were below, within or above, as compared to baseline at Day 0. This outcome presents values for EOS, Hgb and WBC.
Time Frame: At Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 48 | 50
Participants
  EOS, Within-Bellow: number analyzed (Participants) | 48 | 47
  EOS, Within-Bellow | 0 | 0
  EOS, Within-Within: number analyzed (Participants) | 48 | 47
  EOS, Within-Within | 46 | 45
  EOS, Within-Above: number analyzed (Participants) | 48 | 47
  EOS, Within-Above | 2 | 2
  EOS, Above-Below: number analyzed (Participants) | 1 | 4
  EOS, Above-Below | 0 | 0
  EOS, Above-Within: number analyzed (Participants) | 1 | 4
  EOS, Above-Within | 0 | 2
  EOS, Above-Above: number analyzed (Participants) | 1 | 4
  EOS, Above-Above | 1 | 2
  Hgb, Below-Below: number analyzed (Participants) | 1 | 1
  Hgb, Below-Below | 0 | 1
  Hgb, Below-Within: number analyzed (Participants) | 1 | 1
  Hgb, Below-Within | 1 | 0
  Hgb, Below-Above: number analyzed (Participants) | 1 | 1
  Hgb, Below-Above | 0 | 0
  Hgb, Within-Bellow | 1 | 0
  Hgb, Within-Within | 47 | 50
  Hgb, Within-Above | 0 | 0
  WBC, Within-Bellow | 0 | 0
  WBC, Within-Within | 46 | 47
  WBC, Within-Above | 2 | 1
  WBC, Above-Below: number analyzed (Participants) | 1 | 3
  WBC, Above-Below | 0 | 0
  WBC, Above-Within: number analyzed (Participants) | 1 | 3
  WBC, Above-Within | 1 | 2
  WBC, Above-Above: number analyzed (Participants) | 1 | 3
  WBC, Above-Above | 0 | 1

4. Primary Outcome: Number of Subjects With Abnormal Haematological Laboratory Values.
Description: as for outcome 3
Time Frame: At Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 48 | 50
Participants
  EOS, Within-Bellow: number analyzed (Participants) | 48 | 47
  EOS, Within-Bellow | 0 | 0
  EOS, Within-Within: number analyzed (Participants) | 48 | 47
  EOS, Within-Within | 41 | 44
  EOS, Within-Above: number analyzed (Participants) | 48 | 47
  EOS, Within-Above | 7 | 3
  EOS, Above-Below: number analyzed (Participants) | 1 | 4
  EOS, Above-Below | 0 | 0
  EOS, Above-Within: number analyzed (Participants) | 1 | 4
  EOS, Above-Within | 0 | 3
  EOS, Above-Above: number analyzed (Participants) | 1 | 4
  EOS, Above-Above | 1 | 1
  Hgb, Below-Below: number analyzed (Participants) | 1 | 1
  Hgb, Below-Below | 0 | 1
  Hgb, Below-Within: number analyzed (Participants) | 1 | 1
  Hgb, Below-Within | 1 | 0
  Hgb, Below-Above: number analyzed (Participants) | 1 | 1
  Hgb, Below-Above | 0 | 0
  Hgb, Within-Bellow | 0 | 0
  Hgb, Within-Within | 48 | 50
  Hgb, Within-Above | 0 | 0
  WBC, Within-Bellow: number analyzed (Participants) | 48 | 48
  WBC, Within-Bellow | 0 | 1
  WBC, Within-Within: number analyzed (Participants) | 48 | 48
  WBC, Within-Within | 47 | 45
  WBC, Within-Above: number analyzed (Participants) | 48 | 48
  WBC, Within-Above | 1 | 2
  WBC, Above-Below: number analyzed (Participants) | 1 | 3
  WBC, Above-Below | 0 | 0
  WBC, Above-Within: number analyzed (Participants) | 1 | 3
  WBC, Above-Within | 1 | 3
  WBC, Above-Above: number analyzed (Participants) | 1 | 3
  WBC, Above-Above | 0 | 0

5. Primary Outcome: Number of Subjects With Abnormal Haematological Laboratory Values.
Description: Among analysed haematological parameters were eosinophils [EOS], haemoglobin [Hgb], leukocytes (white blood cells) [WBC], lymphocytes [LYM], neutrophils [NEU] and platelets [PLT]. Haematological value ranges assessed were below, within or above, as compared to baseline at Day 0. This outcome presents values for LYM, NEU and PLT
Time Frame: At Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 48 | 50
Participants
  LYM, Below-Below: number analyzed (Participants) | 0 | 2
  LYM, Below-Below | 0 | 0
  LYM, Below-Within: number analyzed (Participants) | 0 | 2
  LYM, Below-Within | 0 | 2
  LYM, Below-Above: number analyzed (Participants) | 0 | 2
  LYM, Below-Above | 0 | 0
  LYM, Within-Bellow: number analyzed (Participants) | 46 | 48
  LYM, Within-Bellow | 1 | 1
  LYM, Within-Within: number analyzed (Participants) | 46 | 48
  LYM, Within-Within | 42 | 45
  LYM, Within-Above: number analyzed (Participants) | 46 | 48
  LYM, Within-Above | 3 | 2
  LYM, Above-Below: number analyzed (Participants) | 3 | 1
  LYM, Above-Below | 0 | 0
  LYM, Above-Within: number analyzed (Participants) | 3 | 1
  LYM, Above-Within | 1 | 1
  LYM, Above-Above: number analyzed (Participants) | 3 | 1
  LYM, Above-Above | 2 | 0
  NEU, Below-Below: number analyzed (Participants) | 1 | 0
  NEU, Below-Below | 0 | 0
  NEU, Below-Within: number analyzed (Participants) | 1 | 0
  NEU, Below-Within | 1 | 0
  NEU, Below-Above: number analyzed (Participants) | 1 | 0
  NEU, Below-Above | 0 | 0
  NEU, Within-Bellow: number analyzed (Participants) | 47 | 48
  NEU, Within-Bellow | 3 | 2
  NEU, Within-Within: number analyzed (Participants) | 47 | 48
  NEU, Within-Within | 44 | 44
  NEU, Within-Above: number analyzed (Participants) | 47 | 48
  NEU, Within-Above | 0 | 2
  NEU, Above-Below: number analyzed (Participants) | 1 | 3
  NEU, Above-Below | 0 | 0
  NEU, Above-Within: number analyzed (Participants) | 1 | 3
  NEU, Above-Within | 0 | 1
  NEU, Above-Above: number analyzed (Participants) | 1 | 3
  NEU, Above-Above | 1 | 2
  PLT, Within-Bellow | 1 | 1
  PLT, Within-Within | 47 | 47
  PLT, Within-Above | 0 | 2
  PLT, Above-Below: number analyzed (Participants) | 1 | 1
  PLT, Above-Below | 0 | 0
  PLT, Above-Within: number analyzed (Participants) | 1 | 1
  PLT, Above-Within | 0 | 0
  PLT, Above-Above: number analyzed (Participants) | 1 | 1
  PLT, Above-Above | 1 | 1

6. Primary Outcome: Number of Subjects With Abnormal Haematological Laboratory Values.
Description: as for outcome 5
Time Frame: At Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 48 | 50
Participants
  LYM, Below-Below: number analyzed (Participants) | 0 | 2
  LYM, Below-Below | 0 | 0
  LYM, Below-Within: number analyzed (Participants) | 0 | 2
  LYM, Below-Within | 0 | 2
  LYM, Below-Above: number analyzed (Participants) | 0 | 2
  LYM, Below-Above | 0 | 0
  LYM, Within-Bellow: number analyzed (Participants) | 46 | 48
  LYM, Within-Bellow | 1 | 0
  LYM, Within-Within: number analyzed (Participants) | 46 | 48
  LYM, Within-Within | 44 | 46
  LYM, Within-Above: number analyzed (Participants) | 46 | 48
  LYM, Within-Above | 1 | 2
  LYM, Above-Below: number analyzed (Participants) | 3 | 1
  LYM, Above-Below | 0 | 0
  LYM, Above-Within: number analyzed (Participants) | 3 | 1
  LYM, Above-Within | 2 | 1
  LYM, Above-Above: number analyzed (Participants) | 3 | 1
  LYM, Above-Above | 1 | 0
  NEU, Below-Below: number analyzed (Participants) | 1 | 0
  NEU, Below-Below | 0 | 0
  NEU, Below-Within: number analyzed (Participants) | 1 | 0
  NEU, Below-Within | 1 | 0
  NEU, Below-Above: number analyzed (Participants) | 1 | 0
  NEU, Below-Above | 0 | 0
  NEU, Within-Bellow: number analyzed (Participants) | 47 | 48
  NEU, Within-Bellow | 0 | 0
  NEU, Within-Within: number analyzed (Participants) | 47 | 48
  NEU, Within-Within | 46 | 48
  NEU, Within-Above: number analyzed (Participants) | 47 | 48
  NEU, Within-Above | 1 | 0
  NEU, Above-Below: number analyzed (Participants) | 1 | 3
  NEU, Above-Below | 0 | 0
  NEU, Above-Within: number analyzed (Participants) | 1 | 3
  NEU, Above-Within | 1 | 3
  NEU, Above-Above: number analyzed (Participants) | 1 | 3
  NEU, Above-Above | 0 | 0
  PLT, Within-Bellow | 1 | 2
  PLT, Within-Within | 47 | 48
  PLT, Within-Above | 0 | 0
  PLT, Above-Below: number analyzed (Participants) | 1 | 1
  PLT, Above-Below | 0 | 0
  PLT, Above-Within: number analyzed (Participants) | 1 | 1
  PLT, Above-Within | 1 | 0
  PLT, Above-Above: number analyzed (Participants) | 1 | 1
  PLT, Above-Above | 0 | 1

7. Primary Outcome: Number of Subjects With Abnormal Biochemical Laboratory Parameter Values by Maximum Grading
Description: Among biochemical parameters tested were ALT, AST and CRE, graded by FDA toxicity grading for biochemistry parameters. Assessed grades were unknown, grade 0 [G0], grade 1 [G1] (mild), grade 2 [G2] (moderate), grade 3 [G3] (severe) and grade 4 [G4] (potentially life threatening), as compared to baseline at Day 0.
Time Frame: From Day 7 up to Day 30
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all subjects with study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  ALT, Unknown-Unknown: number analyzed (Participants) | 0 | 1
  ALT, Unknown-Unknown | 0 | 1
  ALT, Unknown-G0: number analyzed (Participants) | 0 | 1
  ALT, Unknown-G0 | 0 | 0
  ALT, Unknown-G1: number analyzed (Participants) | 0 | 1
  ALT, Unknown-G1 | 0 | 0
  ALT, Unknown-G2: number analyzed (Participants) | 0 | 1
  ALT, Unknown-G2 | 0 | 0
  ALT, Unknown-G3: number analyzed (Participants) | 0 | 1
  ALT, Unknown-G3 | 0 | 0
  ALT, Unknown-G4: number analyzed (Participants) | 0 | 1
  ALT, Unknown-G4 | 0 | 0
  ALT, G0-Unknown: number analyzed (Participants) | 49 | 50
  ALT, G0-Unknown | 0 | 0
  ALT, G0-G0: number analyzed (Participants) | 49 | 50
  ALT, G0-G0 | 48 | 49
  ALT, G0-G1: number analyzed (Participants) | 49 | 50
  ALT, G0-G1 | 1 | 1
  ALT, G0-G2: number analyzed (Participants) | 49 | 50
  ALT, G0-G2 | 0 | 0
  ALT, G0-G3: number analyzed (Participants) | 49 | 50
  ALT, G0-G3 | 0 | 0
  ALT, G0-G4: number analyzed (Participants) | 49 | 50
  ALT, G0-G4 | 0 | 0
  AST, G0-Unknown: number analyzed (Participants) | 48 | 51
  AST, G0-Unknown | 0 | 0
  AST, G0-G0: number analyzed (Participants) | 48 | 51
  AST, G0-G0 | 47 | 49
  AST, G0-G1: number analyzed (Participants) | 48 | 51
  AST, G0-G1 | 1 | 2
  AST, G0-G2: number analyzed (Participants) | 48 | 51
  AST, G0-G2 | 0 | 0
  AST, G0-G3: number analyzed (Participants) | 48 | 51
  AST, G0-G3 | 0 | 0
  AST, G0-G4: number analyzed (Participants) | 48 | 51
  AST, G0-G4 | 0 | 0
  AST, G1-Unknown: number analyzed (Participants) | 1 | 0
  AST, G1-Unknown | 0 | 0
  AST, G1-G0: number analyzed (Participants) | 1 | 0
  AST, G1-G0 | 0 | 0
  AST, G1-G1: number analyzed (Participants) | 1 | 0
  AST, G1-G1 | 1 | 0
  AST, G1-G2: number analyzed (Participants) | 1 | 0
  AST, G1-G2 | 0 | 0
  AST, G1-G3: number analyzed (Participants) | 1 | 0
  AST, G1-G3 | 0 | 0
  AST, G1-G4: number analyzed (Participants) | 1 | 0
  AST, G1-G4 | 0 | 0
  CRE, G0-Unknown | 0 | 0
  CRE, G0-G0 | 49 | 51
  CRE, G0-G1 | 0 | 0
  CRE, G0-G2 | 0 | 0
  CRE, G0-G3 | 0 | 0
  CRE, G0-G4 | 0 | 0

8. Primary Outcome: Number of Subjects With Abnormal Haematological Laboratory Parameter Values by Maximum Grading
Description: Among haematological parameters tested were EOS, decreased Hgb and LYM graded by FDA toxicity grading for haematology parameters. Assessed grades were unknown, grade 0 [G0], grade 1 [G1] (mild), grade 2 [G2] (moderate), grade 3 [G3] (severe) and grade 4 [G4] (potentially life threatening), as compared to baseline at Day 0.
Time Frame: From Day 7 up to Day 30
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  EOS, G0-Unknown | 0 | 0
  EOS, G0-G0 | 48 | 49
  EOS, G0-G1 | 1 | 2
  EOS, G0-G2 | 0 | 0
  EOS, G0-G3 | 0 | 0
  EOS, G0-G4 | 0 | 0
  Hgb/D, G0-Unknown: number analyzed (Participants) | 47 | 49
  Hgb/D, G0-Unknown | 0 | 0
  Hgb/D, G0-G0: number analyzed (Participants) | 47 | 49
  Hgb/D, G0-G0 | 45 | 46
  Hgb/D, G0-G1: number analyzed (Participants) | 47 | 49
  Hgb/D, G0-G1 | 2 | 3
  Hgb/D, G0-G2: number analyzed (Participants) | 47 | 49
  Hgb/D, G0-G2 | 0 | 0
  Hgb/D, G0-G3: number analyzed (Participants) | 47 | 49
  Hgb/D, G0-G3 | 0 | 0
  Hgb/D, G0-G4: number analyzed (Participants) | 47 | 49
  Hgb/D, G0-G4 | 0 | 0
  Hgb/D, G1-Unknown: number analyzed (Participants) | 2 | 1
  Hgb/D, G1-Unknown | 0 | 0
  Hgb/D, G1-G0: number analyzed (Participants) | 2 | 1
  Hgb/D, G1-G0 | 0 | 1
  Hgb/D, G1-G1: number analyzed (Participants) | 2 | 1
  Hgb/D, G1-G1 | 2 | 0
  Hgb/D, G1-G2: number analyzed (Participants) | 2 | 1
  Hgb/D, G1-G2 | 0 | 0
  Hgb/D, G1-G3: number analyzed (Participants) | 2 | 1
  Hgb/D, G1-G3 | 0 | 0
  Hgb/D, G1-G4: number analyzed (Participants) | 2 | 1
  Hgb/D, G1-G4 | 0 | 0
  Hgb/D, G4-Unknown: number analyzed (Participants) | 0 | 1
  Hgb/D, G4-Unknown | 0 | 0
  Hgb/D, G4-G0: number analyzed (Participants) | 0 | 1
  Hgb/D, G4-G0 | 0 | 0
  Hgb/D, G4-G1: number analyzed (Participants) | 0 | 1
  Hgb/D, G4-G1 | 0 | 0
  Hgb/D, G4-G2: number analyzed (Participants) | 0 | 1
  Hgb/D, G4-G2 | 0 | 0
  Hgb/D, G4-G3: number analyzed (Participants) | 0 | 1
  Hgb/D, G4-G3 | 0 | 0
  Hgb/D, G4-G4: number analyzed (Participants) | 0 | 1
  Hgb/D, G4-G4 | 0 | 1
  LYM, G0-Unknown | 0 | 0
  LYM, G0-G0 | 49 | 48
  LYM, G0-G1 | 0 | 2
  LYM, G0-G2 | 0 | 1
  LYM, G0-G3 | 0 | 0
  LYM, G0-G4 | 0 | 0

9. Primary Outcome: Number of Subjects With Abnormal Haematological Laboratory Parameter Values by Maximum Grading
Description: Among haematological parameters tested were NEU, PLT, decreased WBC and increased WBC/I, graded by FDA toxicity grading for haematology parameters. Assessed grades were unknown, grade 0 [G0], grade 1 [G1] (mild), grade 2 [G2] (moderate), grade 3 [G3] (severe) and grade 4 [G4] (potentially life threatening), as compared to baseline at Day 0.
Time Frame: From Day 7 up to Day 30
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  NEU, G0-Unknown: number analyzed (Participants) | 47 | 49
  NEU, G0-Unknown | 0 | 0
  NEU, G0-G0: number analyzed (Participants) | 47 | 49
  NEU, G0-G0 | 46 | 47
  NEU, G0-G1: number analyzed (Participants) | 47 | 49
  NEU, G0-G1 | 1 | 2
  NEU, G0-G2: number analyzed (Participants) | 47 | 49
  NEU, G0-G2 | 0 | 0
  NEU, G0-G3: number analyzed (Participants) | 47 | 49
  NEU, G0-G3 | 0 | 0
  NEU, G0-G4: number analyzed (Participants) | 47 | 49
  NEU, G0-G4 | 0 | 0
  NEU, G1-Unknown: number analyzed (Participants) | 2 | 2
  NEU, G1-Unknown | 0 | 0
  NEU, G1-G0: number analyzed (Participants) | 2 | 2
  NEU, G1-G0 | 0 | 2
  NEU, G1-G1: number analyzed (Participants) | 2 | 2
  NEU, G1-G1 | 1 | 0
  NEU, G1-G2: number analyzed (Participants) | 2 | 2
  NEU, G1-G2 | 1 | 0
  NEU, G1-G3: number analyzed (Participants) | 2 | 2
  NEU, G1-G3 | 0 | 0
  NEU, G1-G4: number analyzed (Participants) | 2 | 2
  NEU, G1-G4 | 0 | 0
  PLT, G0-Unknown | 0 | 0
  PLT, G0-G0 | 49 | 49
  PLT, G0-G1 | 0 | 2
  PLT, G0-G2 | 0 | 0
  PLT, G0-G3 | 0 | 0
  PLT, G0-G4 | 0 | 0
  WBC/D, G0-Unknown | 0 | 0
  WBC/D, G0-G0 | 49 | 50
  WBC/D, G0-G1 | 0 | 1
  WBC/D, G0-G2 | 0 | 0
  WBC/D, G0-G3 | 0 | 0
  WBC/D, G0-G4 | 0 | 0
  WBC/I, G0-Unknown: number analyzed (Participants) | 49 | 50
  WBC/I, G0-Unknown | 0 | 0
  WBC/I, G0-G0: number analyzed (Participants) | 49 | 50
  WBC/I, G0-G0 | 47 | 49
  WBC/I, G0-G1: number analyzed (Participants) | 49 | 50
  WBC/I, G0-G1 | 2 | 1
  WBC/I, G0-G2: number analyzed (Participants) | 49 | 50
  WBC/I, G0-G2 | 0 | 0
  WBC/I, G0-G3: number analyzed (Participants) | 49 | 50
  WBC/I, G0-G3 | 0 | 0
  WBC/I, G0-G4: number analyzed (Participants) | 49 | 50
  WBC/I, G0-G4 | 0 | 0
  WBC/I, G1-Unknown: number analyzed (Participants) | 0 | 1
  WBC/I, G1-Unknown | 0 | 0
  WBC/I, G1-G0: number analyzed (Participants) | 0 | 1
  WBC/I, G1-G0 | 0 | 1
  WBC/I, G1-G1: number analyzed (Participants) | 0 | 1
  WBC/I, G1-G1 | 0 | 0
  WBC/I, G1-G2: number analyzed (Participants) | 0 | 1
  WBC/I, G1-G2 | 0 | 0
  WBC/I, G1-G3: number analyzed (Participants) | 0 | 1
  WBC/I, G1-G3 | 0 | 0
  WBC/I, G1-G4: number analyzed (Participants) | 0 | 1
  WBC/I, G1-G4 | 0 | 0

10. Primary Outcome: Number of Subjects With Haematology Change From Baseline by Maximum Grade
Description: Assessed laboratory parameter changed from baseline was haemoglobin (Hgb). FDA grading for Hgb (change from baseline) was not applicable a baseline.
Time Frame: From Day 7 up to Day 30
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  Hgb, G0 | 15 | 15
  Hgb, G1 | 34 | 35
  Hgb, G2 | 0 | 1
  Hgb, G3 | 0 | 0
  Hgb, G4 | 0 | 0

11. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimetres (mm) of injection site. All solicited local symptoms are considered as related to the vaccination.
Time Frame: During a 7-day follow-up period (from Day 0 to Day 6) after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  Any Pain | 27 | 46
  Grade 3 Pain | 1 | 1
  Any Redness | 0 | 1
  Grade 3 Redness | 0 | 1
  Any Swelling | 0 | 1
  Grade 3 Swelling | 0 | 0

12. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, temperature (defined as oral temperature equal to or above [≥] 37.5 degrees Celsius [°C] for oral, axillary or tympanic route), gastrointestinal symptoms (gastro) including nausea, vomiting, diarrhoea and/or abdominal pain; and headache. Any = occurrence of the symptom regardless of intensity grade and relationship to the vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During a 7-day follow-up period (from Day 0 to Day 6) after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants
  Any Fatigue | 20 | 23
  Grade 3 Fatigue | 4 | 1
  Related Fatigue | 15 | 15
  Any Gastro. | 14 | 14
  Grade 3 Gastro. | 2 | 1
  Related Gastro. | 8 | 9
  Any Headache | 14 | 17
  Grade 3 Headache | 3 | 1
  Related Headache | 5 | 9
  Any temperature | 2 | 2
  Grade 3 Temperature | 0 | 0
  Related temperature | 0 | 2

13. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During a 30-day follow-up period (from Day 0 to Day 29) after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants | 23 | 28

14. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From vaccination (Day 0) up to study end (Day 30)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Group | Boostrix Group
Number analyzed (Participants) | 49 | 51
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs during the 30-Day follow-up period after vaccination; SAEs from Day 0 up to study end Day 30.
Arm/Group | GSK3003891A Group | Boostrix Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 27/49 | 46/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3003891A Group (N=49) | Boostrix Group (N=51)
Gastrointestinal disorder (Gastrointestinal disorders) | 14 (15) | 14 (14)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Fatigue (General disorders) | 20 (20) | 24 (27)
Pain (General disorders) | 27 (27) | 46 (46)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 18 (21) | 25 (29)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.